CLINICAL TRIAL: NCT02750891
Title: A Phase 1/2 Study of DSP-7888 in Pediatric Patients With Relapsed or Refractory High Grade Gliomas
Brief Title: A Study of DSP-7888 in Pediatric Patients With Relapsed or Refractory High Grade Gliomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DB601001; JapicCTI-163216 (Registry Identifier: JAPIC Clinical Trials Information)
Record Dates: First submitted 2016-04-13; First posted 2016-04-26 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Glioblastoma; Diffuse Intrinsic Pontine Glioma
Keywords: high grade glioma; HGG; DIPG
MeSH Terms: conditions — Glioblastoma; Diffuse Intrinsic Pontine Glioma; Glioma

ARMS (1):
- DSP-7888 (Experimental)
  Interventions: Drug: DSP-7888

INTERVENTIONS:
Drug: DSP-7888 — Phase1 portion: 1.75 or 3.5 mg/body, Id every 1-4 weeks Phase 2 portion: recommended phase 2 dose, Id every 1-4 weeks

SUMMARY:
This is a phase 1/2, uncontrolled, open-label, multicenter study in patients with recurrent and relapsed diffuse intrinsic pontine glioma, glioblastoma, or grade III or IV glioma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meeting any of the conditions a) to c) below:

   1. Have a diagnosis of diffuse intrinsic pontine glioma on the basis of imaging findings on magnetic resonance imaging (MRI) and clinical course
   2. Have histologically or cytologically confirmed glioblastoma
   3. Not meeting a) and b) above, but have histologically or cytologically confirmed grade III or IV glioma
2. Patients who will be able to be hospitalized from the initial dose of DSP-7888 until the end of the post-initial dose observation (In Phase 1 part only, patients may be permitted to have a temporary overnight leave during the hospitalization.)
3. Patients aged < 20 years at the time of informed consent
4. Patients for whom either the legally acceptable representative or the patient (if aged ≥ 16 years) have provided written voluntary consent to participation in this study after fully receiving and understanding the information about this study, including study objectives, contents, expected pharmacological actions and effects, and foreseeable risks
5. Patients for whom standard therapy failed or no standard therapy is established
6. Diffuse intrinsic pontine glioma patients must received radiotherapy-based treatment or chemotherapy (if radiotherapy is not indicated) at least one cycle and subsequently had tumor enlargement accompanied by tumor-related symptomatic worsening (except for worsening due to dose reduction of steroid therapy for brain edema)
7. Glioblastoma patients and grade III or IV glioma patients must had radiologically evident tumor re-enlargement or recurrence
8. Patients with an ECOG PS score of 0 to 2 at enrollment. Patients with a PS score of 3 or 4 due to neurological symptoms associated with the primary disease may be eligible if appropriate in the opinion of the investigator or subinvestigator.
9. Patients with a life expectancy of 2 months (60 days)
10. Patients with a HLA type of HLA-A*24:02 or A*02:01/06
11. Patients with adequate major organ functions meeting the following criteria on the basis of laboratory data within 28 days before enrollment:

    Neutrophil count: 1000/μL Platelet count: 5.0 ×104/μL Hemoglobin: 9.0 g/dL Serum creatinine: 2-fold the upper limit of the normal range of the study site (ULN) Total bilirubin: 2-fold the ULN AST, ALT: 3-fold the ULN
12. Female patients of childbearing potential must have a negative pregnancy test within 4 weeks (28 days) before enrollment
13. Female patients of childbearing potential and male patients with female partners of childbearing potential must agree to use appropriate contraception from the time of consent until 180 days after the last dose of the study drug to avoid pregnancy

Exclusion Criteria:

1. Patients with grade 3 infection according to the CTCAE v4.0
2. Patients with a positive test result for HIV antibody, HBs antigen, or HCV antibody
3. Patients with multiple or disseminated primary lesions (Multiple nodules in the same tumor cavity will be acceptable.)
4. Patients with other malignancies
5. Patients with significant diseases at enrollment that may affect study treatment, such as New York Heart Association (NYHA) Functional Class III or IV heart disease, CTCAE v4.0 grade 3 arrhythmia, angina pectoris, abnormal electrocardiogram findings, interstitial pneumonia or pulmonary fibrosis
6. Patients with uncontrollable complications
7. Patients who underwent allogeneic hematopoietic stem cell transplant
8. Patients who received any of the following treatments within the specified period before enrollment

   * Nitrosoureas, mitomycin C: <42 days
   * Chemotherapy (including molecular-targeted drugs), radiotherapy: <21 days
   * Surgery, blood transfusion, erythropoiesis-stimulating drugs, endocrine therapy, immunotherapy (including biological response modifier [BRM] therapy): <14 days
9. Pregnant or breastfeeding women
10. Patients with concurrent autoimmune disease or a history of chronic or recurrent autoimmune disease, or patients who require long-term systemic steroid therapy (excluding therapy given on a PRN basis). However, steroid therapy for brain edema (prednisolone-equivalent dose of 30 mg/m2) and steroid replacement therapy at a physiologic dose will be acceptable.
11. Patients with any ongoing CTCAE v4.0 grade 2 adverse effects of prior treatment (excluding alopecia and phlebitis)
12. Patients who received any other investigational product or post-marketing study drug within 4 weeks (28 days) before enrollment
13. Patients with a history of allergy to any oil-based agents
14. Patients who previously received DSP-7888-containing WT1 peptide, or WT1 immunotherapy
15. Patients who are inappropriate for participation in the study for other reasons in the opinion of the investigator or subinvestigator

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
DLT (dose-limiting toxicity) | 4 weeks
  Safety and tolerability assessed by dose-limiting toxicity (DLT)
Overall Survival （OS） | 24 months
  Participants follow-up for overall survival will occur. Maximum follow-up time is 2 year after the initial administration of the last subject.

SECONDARY OUTCOMES:
Overall Response Rate（ORR） | 6 months
  Antitumor effect as assessed according to the Response Assessment in Neuro-Oncology (RANO) criteria
Progression-free survival (PFS) | 6 months
adverse events (AEs) | 12 months
  Safety and tolerability assessed by adverse events (AEs)
serious adverse events (SAEs) | 12 months
  Safety and tolerability assessed by serious adverse events (SAEs)
DTH （delayed-type hypersensitivity） | 6 months
  Explore efficacy related biomarkers assessed by delayed-type hypersensitivity (DTH) reactions to WT1 peptide
WT1 peptide-specific CTL-induction activity | 6 months
  Explore efficacy related biomarkers assessed by WT1 peptide-specific CTL-induction activity.
expression of WT1 in biopsy tissues | 6 months
  Explore efficacy related biomarkers assessed in biopsy tissues
expression of HLA in biopsy tissues | 6 months
  Explore efficacy related biomarkers assessed in biopsy tissues
expression of PD-L1 in biopsy tissues | 6 months
  Explore efficacy related biomarkers assessed in biopsy tissues

CONTACTS AND LOCATIONS:
Overall Officials: Sumitomo Pharma Co., Ltd. Japan, Study Director — Sumitomo Pharma Co., Ltd.
Locations (6):
- Japan (6):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Kanagawa Children's Medical Center, Yokohama, Kanagawa
  - Osaka University Hospital, Suita, Osaka
  - National Center for Child Health and Development, Setagaya City, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - Osaka City General Hospital, Osaka